CLINICAL TRIAL: NCT03408899
Title: A Phase 1 Safety and Pharmacokinetic Study of PC-1005 (MIV-150/Zinc Acetate/Carrageenan Gel) Administered Rectally to HIV-1 Seronegative Adults
Brief Title: Evaluating the Safety and Pharmacokinetics of PC-1005 Administered Rectally to HIV-1 Seronegative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MTN-037; 35122 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections
Keywords: Microbicides
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PC-1005 (Experimental): All participants will receive 3 single escalating doses of PC-1005 gel during Visits 3, 5, and 7, with a 2-to-6-week washout period between dosing visits. Each participant will be on study for approximately 3 to 5 months.
  Interventions: Drug: PC-1005 gel

INTERVENTIONS:
Drug: PC-1005 gel — PC-1005 (0.002% MIV-150/0.3% zinc acetate in 3.0% carrageenan gel) in 4 mL, 16 mL, and 32 mL doses administered rectally.

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of PC-1005 gel when used as a rectal microbicide in HIV-uninfected men and women (cis or transgender) with a history of consensual receptive anal intercourse.

DETAILED DESCRIPTION:
PC-1005 is a multipurpose prevention technology (MPT) microbicide in development that is active against HIV, HPV, and HSV-2. This study will evaluate the safety and pharmacokinetics of PC-1005 gel when administered rectally.

The study will enroll HIV-uninfected men and women (cis or transgender) with a history of consensual receptive anal intercourse. All participants will receive 3 single escalating doses of rectally administered PC-1005: 4 mL, 16 mL and 32 mL.

The study includes a total of 9 clinic visits and 1 follow-up contact by phone or in person. Participants will receive doses of PC-1005 at Visits 3, 5, and 7. A 2-to-6 week washout period will follow each dosing visit. If no adverse events that preclude continuation to the next dose are identified during this period, participants will receive the next scheduled dose of PC-1005. Participation in this study will last approximately 3 to 5 months.

Study visits will include physical examinations, throat swabs, behavioral assessments and interviews, and collection of blood, urine, rectal tissue, and cervical, vaginal, and rectal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (cis or transgender) who are 18 years or older at Screening, verified per site standard operating procedure (SOP)
* Able and willing to provide written informed consent
* HIV-1/2 uninfected at Screening and Enrollment, per applicable algorithm in the protocol and willing to receive HIV test results
* Able and willing to provide adequate locator information, as defined in site SOP
* Available to return for all study visits and willing to comply with study participation requirements
* In general good health at Screening and Enrollment, as determined by the site Investigator of Record (IoR) or designee
* At Screening, history of consensual receptive anal intercourse (RAI) at least once in their lifetime per participant report
* Willing to not take part in other research studies involving drugs, medical devices, genital or rectal products, or vaccines for the duration of study participation (including the time between Screening and Enrollment)
* Willing to follow abstinence requirements for the duration of study participation (See the protocol for additional information)
* For participants of childbearing potential: a negative pregnancy test at Screening and Enrollment
* For participants of childbearing potential: Per participant report at Enrollment, using an effective method of contraception and intending to use an effective method for the duration of study participation; these include:

  * Hormonal methods, excluding vaginal rings
  * Intrauterine device (IUD) inserted at least 42 days prior to Enrollment (but not past the maximum length of recommended usage according to package instructions)
  * Sterilization of participant or partner at least 42 days prior to Enrollment
  * Self-identifies as having sex with women exclusively

Exclusion Criteria:

* At Screening:

  * Hemoglobin Grade 1 or higher*
  * Platelet count Grade 1 or higher*
  * White blood count Grade 2 or higher*
  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) Grade 1 or higher*
  * Serum creatinine greater than 1.3x the site laboratory upper limit of normal (ULN)
  * International normalized ratio (INR) greater than 1.5x the site laboratory ULN
  * History of inflammatory bowel disease by participant report
  * * As per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1, July 2017
  * Note: Otherwise eligible participants with an exclusionary test result can be re-tested during the screening process. If a participant is re-tested and a non-exclusionary result is documented within 45 days of providing informed consent for screening, the participant may be enrolled.
* Known adverse reaction to latex or polyurethane (ever)
* Anticipated use of and/or unwillingness to abstain from the following medications during study participation:

  * Anticoagulant medications
  * Rectally-administered medications
* Known adverse reaction to any of the components of the study product
* Use of pre-exposure prophylaxis (PrEP) for HIV prevention within 1 month prior to Enrollment, and/or anticipated use and/or unwillingness to abstain from PrEP during trial participation
* Use of post-exposure prophylaxis (PEP) for potential HIV exposure within the 3 months prior to Enrollment
* Condomless RAI and/or penile-vaginal intercourse with a partner who is known to be HIV-positive or whose status is unknown in the 6 months prior to Enrollment
* Non-therapeutic injection drug use in the 12 months prior to Enrollment
* Participation in research studies involving drugs, medical devices, genital or rectal products, or vaccines within 30 days of the Enrollment Visit
* Gynecologic, genital, or rectal procedure (e.g., tubal ligation, dilation and curettage, piercing, hemorrhoidal resection, polyp removal) 60 days or less prior to Enrollment, or rectal biopsy, 7 days or less prior to Enrollment. Note: Colposcopy and cervical biopsies for evaluation of an abnormal Pap test as well as IUD insertion/removal are not exclusionary. Anoscopy and endoscopy without rectal biopsies are not exclusionary
* Per participant report, medical records, clinical diagnosis and/or diagnostic testing at either Screening or Enrollment:

  * Diagnosis or treatment of any anogenital sexually transmitted infection (STI) in the past 3 months (including window between Screening and Enrollment)
  * Symptoms, clinical or laboratory diagnosis of active pharyngeal, anorectal infection or reproductive tract infection (RTI) requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines (http://www.cdc.gov/std/treatment)
  * Current symptomatic urinary tract infection (UTI)
  * Infections requiring treatment include Neisseria gonorrhea (GC), Chlamydia trachomatis (CT) infection, syphilis, active herpes simplex virus (HSV) lesions, anogenital sores or ulcers, or symptomatic genital warts, chancroid, pelvic inflammatory disease (PID), symptomatic bacterial vaginosis (BV), symptomatic vaginal candidiasis, other vaginitis, and trichomoniasis.
  * Note: Otherwise eligible participants with an exclusionary UTI, BV and/or candida finding may be re-tested during the screening process.
  * Note: HSV-1 or HSV-2 seropositive diagnosis with no active lesions is permitted since treatment is not required.
* Participants who meet any of the following additional criteria will be excluded from the study:

  * Pregnant or breastfeeding at either Screening or Enrollment or planning to become pregnant or begin breastfeeding during study participation. Note: A documented negative pregnancy test performed by study staff is required for inclusion; however, a self-reported pregnancy is adequate for exclusion from screening/enrollment into the study.
  * Last pregnancy outcome 90 days or less prior to Screening
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Study Chair — Johns Hopkins University
Locations (2):
- United States (2):
  - Alabama CRS, Birmingham, Alabama
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Ho K, Hoesley C, Anderson PL, Fernandez-Romero JA, Friedland BA, Kelly CW, Jiao Y, Edick S, Brand R, Kunjara Na Ayudhya RP, Zyhowski A, Hartman DJ, Reddy NB, Al-Khouja A, Piper J, Bauermeister JA, Teleshova N, Melo C, Cornejal N, Barnable P, Singh D, Scheckter R, McClure T, Hillier SL, Hendrix CW; MTN-037 Study Team. Phase I Dose Volume Escalation of Rectally Administered PC-1005 to Assess Safety, Pharmacokinetics, and Antiviral Pharmacodynamics as a Multipurpose Prevention Technology (MTN-037). J Acquir Immune Defic Syndr. 2024 Dec 1;97(4):379-386. doi: 10.1097/QAI.0000000000003506. PMID 39808074

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant terminated early due to "Lost to follow-up". One additional participant enrolled as replacement. Thus a total of 13 participants enrolled in the study.
Groups:
- All Enrolled Participants: All enrolled participants will receive PC-1005 Gel in 4mL, 16mL, and 32mL dose.
Period: PC-1005 Gel: 4 mL Dose
Arm/Group | All Enrolled Participants
Started | 13
Completed | 12
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: PC-1005 Gel: 16 mL Dose
Arm/Group | All Enrolled Participants
Started | 12
Completed | 12
Not Completed | 0
Period: PC-1005 Gel: 32 mL Dose
Arm/Group | All Enrolled Participants
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PC-1005
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 33.1 [28 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 6
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Height [Mean (Inter-Quartile Range); unit: cm] | 171.0 [162.6 to 177.8]
Weight [Mean (Inter-Quartile Range); unit: kg] | 94.3 [80.3 to 114]
BMI [Mean (Inter-Quartile Range); unit: kg/m^2] | 32.1 [27.5 to 35.1]

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Grade 2 or Higher Adverse Events (AEs)
Description: AEs are defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 and/or Addenda 1, 2 and 3 (Female Genital [Dated November 2007], Male Genital [Dated November 2007] and Rectal [Clarification Dated May 2012] Grading Tables for Use in Microbicide Studies).
Time Frame: Measured through participants' last study visit which will occur at Month 3 to 5, depending on the participant
Measure: Count of Participants; unit: Participants
Groups:
- 4 mL: All participants who received 4 mL of PC-1005 gel at Visits 3.
  PC-1005 gel: PC-1005 (0.002% MIV-150/0.3% zinc acetate in 3.0% carrageenan gel) in 4 mL dose administered rectally.
- 16 mL: All participants who received 16 mL of PC-1005 gel at Visits 5.
  PC-1005 gel: PC-1005 (0.002% MIV-150/0.3% zinc acetate in 3.0% carrageenan gel) in 16 mL dose administered rectally.
- 32 mL: All participants who received 32 mL of PC-1005 gel at Visits 7.
  PC-1005 gel: PC-1005 (0.002% MIV-150/0.3% zinc acetate in 3.0% carrageenan gel) in 32 mL dose administered rectally.
Arm/Group | 4 mL | 16 mL | 32 mL
Number analyzed (Participants) | 13 | 12 | 12
Participants | 1 | 2 | 0

2. Primary Outcome: MIV-150 Concentrations in Plasma
Description: Descriptive statistics such as the mean and median and corresponding 95% confidence intervals will be used to describe the MIV-150 concentrations in all biological matrices assessed at all scheduled time points
Time Frame: Measured through participants' last study visit which will occur at Month 3 to 5, depending on the participant
Population: Participants are randomly assigned 1:1:1 to provide samples of rectal fluid 48 hours after one of the three dose administrations.
  One participant missed 2 hour postdosing plasma sample collection at 4mL dosing visit.
  One participant missed 1 hour postdosing plasma sample collection at 16mL dosing visit.
  One participant missed 24 hour postdosing plasma sample collection at 32mL dosing visit.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 4 mL | 16 mL | 32 mL
Number analyzed (Participants) | 13 | 12 | 12
pg/mL
  Predosing | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  1 hour postdosing: number analyzed (Participants) | 13 | 11 | 12
  1 hour postdosing | 74.0 [52.0 to 86.0] | 164.0 [87.0 to 187.0] | 158.5 [110.0 to 267.5]
  2 hours postdosing: number analyzed (Participants) | 12 | 12 | 12
  2 hours postdosing | 66.5 [45.0 to 83.5] | 183.5 [162.0 to 211.0] | 171.0 [98.0 to 316.0]
  3 hours postdosing | 37.0 [23.0 to 54.0] | 134.0 [84.0 to 191.5] | 143.0 [66.0 to 172.5]
  4 hours postdosing | 24.0 [13.0 to 48.0] | 86.5 [63.0 to 143.5] | 105.0 [40.0 to 138.5]
  5-6 hours postdosing | 13.0 [11.0 to 28.0] | 57.0 [42.5 to 88.0] | 63.5 [25.0 to 121.0]
  24 hours postdosing: number analyzed (Participants) | 13 | 12 | 11
  24 hours postdosing | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 22.0]
  48 hours postdosing: number analyzed (Participants) | 4 | 4 | 4
  48 hours postdosing | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

3. Primary Outcome: MIV-150 Concentrations in Rectal Fluid
Description: as for outcome 2
Time Frame: Measured through participants' last study visit which will occur at Month 3 to 5, depending on the participant
Population: Participants are randomized 1:1:1:1 to provide samples of rectal fluid in one of the following time periods after dose administration : 0.5-1 hour; 1.5-3 hours; 3.5-5 hours, or 24 hours.
  Participants are randomly assigned 1:1:1 to provide samples of rectal fluid 48 hours after one of the three dose administrations.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | 4 mL | 16 mL | 32 mL
Number analyzed (Participants) | 13 | 12 | 12
ng/mL
  0.5-1 hour postdosing: number analyzed (Participants) | 3 | 3 | 3
  0.5-1 hour postdosing | 122.0 [13.2 to 11464.0] | 135.0 [20.2 to 3691.0] | 104.0 [72.8 to 7854.0]
  1.5-3 hour postdosing: number analyzed (Participants) | 4 | 3 | 3
  1.5-3 hour postdosing | 19.3 [14.1 to 41.9] | 23.2 [10.8 to 420.0] | 4582.0 [116.0 to 7272.0]
  3.5-5 hour postdosing: number analyzed (Participants) | 3 | 3 | 3
  3.5-5 hour postdosing | 19.6 [7.8 to 66.7] | 14.9 [3.1 to 37.0] | 39.7 [4.8 to 419.0]
  24 hour postdosing: number analyzed (Participants) | 3 | 3 | 3
  24 hour postdosing | 0 [0 to 0] | 5.9 [2.5 to 6.8] | 0 [0 to 131.0]
  48 hour postdosing: number analyzed (Participants) | 4 | 4 | 4
  48 hour postdosing | 0 [0 to 0] | 0 [0 to 16.9] | 0 [0 to 0]

4. Primary Outcome: MIV-150 Concentrations in Rectal Mucosal Tissue Homogenates
Description: as for outcome 2
Time Frame: Measured through participants' last study visit which will occur at Month 3 to 5, depending on the participant
Population: Three participants are randomized to provide rectal tissue sample in one of the following time periods after dose administration : 0.5-1 hour; 1.5-3 hours; 3.5-5 hours, or 24 hours.
  Four participants are randomized to provide rectal tissue sample 48 hours after each of the three dose administrations.
  Two participants had late sample at 4mL dose.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | 4 mL | 16 mL | 32 mL
Number analyzed (Participants) | 13 | 12 | 12
ng/mL
  0.5-1 hour postdosing: number analyzed (Participants) | 2 | 3 | 3
  0.5-1 hour postdosing | 1.4 [0.8 to 1.9] | 46.0 [30.7 to 831.0] | 79.7 [11.9 to 116.0]
  1.5-3 hour postdosing: number analyzed (Participants) | 4 | 3 | 3
  1.5-3 hour postdosing | 0 [0 to 3.6] | 12.7 [4.8 to 313.0] | 35.8 [2.5 to 186.0]
  3.5-5 hour postdosing: number analyzed (Participants) | 4 | 3 | 3
  3.5-5 hour postdosing | 0 [0 to 0.9] | 4.8 [0 to 6.5] | 0 [0 to 0]
  24 hour postdosing: number analyzed (Participants) | 3 | 3 | 3
  24 hour postdosing | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  48 hour postdosing: number analyzed (Participants) | 4 | 4 | 4
  48 hour postdosing | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Participant Self-report Gel Acceptability - Ease of Use
Description: Response for "Overall, how easy or difficult was it to use the gel when applied by clinic staff?" at exit self-interview questionnaire.
Time Frame: Through study completion, approximately 3-5 months for each participant
Measure: Count of Participants; unit: Participants
Groups:
- Overall: All participants who completed the exit self-interview questionnaire
Arm/Group | Overall
Number analyzed (Participants) | 12
Participants
  Very difficult | 0
  Difficult | 0
  Easy | 3
  Very Easy | 9

6. Secondary Outcome: Participant Self-report Gel Acceptability - Feeling When Inserted
Description: Response for "Overall, how did it feel to have the gel inside you?" at exit self-interview questionnaire.
Time Frame: Through study completion, approximately 3-5 months for each participant
Population: All participants who completed the exit self-interview questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 12
Participants
  Very comfortable | 2
  Comfortable | 8
  Uncomfortable | 1
  Very uncomfortable | 1

7. Secondary Outcome: Participant Self-report Gel Acceptability - Problems With Gel Use
Description: Responses for questions related to problem with gel use at exit self-interview questionnaire
Time Frame: Through study completion, approximately 3-5 months for each participant
Population: All participants who completed the exit self-interview questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 12
Participants
  Did you have any problems using this product?: Yes | 0
  Did you have any problems using this product?: No | 12
  Did you experience any leakage after you used the product?: Yes | 2
  Did you experience any leakage after you used the product?: No | 10
  Did you experience any soiling of your underwear or linens from the gel?: Yes | 0
  Did you experience any soiling of your underwear or linens from the gel?: No | 12
  Did you experience any diarrhea after using the gel?: Yes | 0
  Did you experience any diarrhea after using the gel?: No | 12
  Did you experience any other stomach or abdominal problems after using the gel?: Yes | 2
  Did you experience any other stomach or abdominal problems after using the gel?: No | 10
  Did you experience any any dryness after using the product?: Yes | 0
  Did you experience any any dryness after using the product?: No | 12

8. Secondary Outcome: Participant Self-report Gel Acceptability - Gel Acceptability
Description: Response for questions related to gel acceptability at exit self-interview questionnaire.
Time Frame: Through study completion, approximately 3-5 months for each participant
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 12
Participants
  Overall, how much did you like the gel?: 1 (Dislike very much) | 0
  Overall, how much did you like the gel?: 2 | 0
  Overall, how much did you like the gel?: 3 | 0
  Overall, how much did you like the gel?: 4 | 1
  Overall, how much did you like the gel?: 5 | 3
  Overall, how much did you like the gel?: 6 | 0
  Overall, how much did you like the gel?: 7 | 2
  Overall, how much did you like the gel?: 8 | 3
  Overall, how much did you like the gel?: 9 | 1
  Overall, how much did you like the gel?: 10 (Like very much) | 2
  Overall, how much did you like the gel?: Not Applicable | 0
  How much did you like the smell of the gel?: 1 (Dislike very much) | 0
  How much did you like the smell of the gel?: 2 | 0
  How much did you like the smell of the gel?: 3 | 0
  How much did you like the smell of the gel?: 4 | 1
  How much did you like the smell of the gel?: 5 | 0
  How much did you like the smell of the gel?: 6 | 1
  How much did you like the smell of the gel?: 7 | 0
  How much did you like the smell of the gel?: 8 | 0
  How much did you like the smell of the gel?: 9 | 0
  How much did you like the smell of the gel?: 10 (Like very much) | 0
  How much did you like the smell of the gel?: Not Applicable | 10
  How much did you like the consistency of the gel?: 1 (Dislike very much) | 0
  How much did you like the consistency of the gel?: 2 | 0
  How much did you like the consistency of the gel?: 3 | 0
  How much did you like the consistency of the gel?: 4 | 1
  How much did you like the consistency of the gel?: 5 | 1
  How much did you like the consistency of the gel?: 6 | 2
  How much did you like the consistency of the gel?: 7 | 1
  How much did you like the consistency of the gel?: 8 | 2
  How much did you like the consistency of the gel?: 9 | 3
  How much did you like the consistency of the gel?: 10 (Like very much) | 2
  How much did you like the consistency of the gel?: Not Applicable | 0
  How much did you like how the gel felt inside your rectum immediately after inserting it?: 1 (Dislike very much) | 0
  How much did you like how the gel felt inside your rectum immediately after inserting it?: 2 | 0
  How much did you like how the gel felt inside your rectum immediately after inserting it?: 3 | 1
  How much did you like how the gel felt inside your rectum immediately after inserting it?: 4 | 0
  How much did you like how the gel felt inside your rectum immediately after inserting it?: 5 | 2
  How much did you like how the gel felt inside your rectum immediately after inserting it?: 6 | 2
  How much did you like how the gel felt inside your rectum immediately after inserting it?: 7 | 2
  How much did you like how the gel felt inside your rectum immediately after inserting it?: 8 | 2
  How much did you like how the gel felt inside your rectum immediately after inserting it?: 9 | 2
  How much did you like how the gel felt inside your rectum immediately after inserting it?: 10 (Like very much) | 1
  How much did you like how the gel felt inside your rectum immediately after inserting it?: Not Applicable | 0
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: 1 (Dislike very much) | 0
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: 2 | 0
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: 3 | 0
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: 4 | 1
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: 5 | 3
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: 6 | 2
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: 7 | 1
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: 8 | 1
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: 9 | 2
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: 10 (Like very much) | 2
  How much did you like how the gel felt inside your rectum 30 minutes after inserting it?: Not Applicable | 0

9. Secondary Outcome: MIV-150 Concentrations in Vaginal Fluid
Description: as for outcome 2
Time Frame: Measured through participants' last study visit which will occur at Month 3 to 5, depending on the participant
Population: Participants are randomized 1:1:1:1 to provide samples of rectal fluid in one of the following time periods after dose administration : 0.5-1 hour; 1.5-3 hours; 3.5-5 hours, or 24 hours.
  Participants are randomly assigned 1:1:1 to provide samples of rectal fluid 48 hours after one of the three dose administrations.
  Female participants only.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | 4 mL | 16 mL | 32 mL
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  0.5-1 hour postdosing: number analyzed (Participants) | 1 | 1 | 1
  0.5-1 hour postdosing | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  1.5-3 hour postdosing: number analyzed (Participants) | 1 | 1 | 1
  1.5-3 hour postdosing | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  3.5-5 hour postdosing: number analyzed (Participants) | 2 | 1 | 2
  3.5-5 hour postdosing | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  24 hour postdosing: number analyzed (Participants) | 2 | 1 | 2
  24 hour postdosing | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  48 hour postdosing: number analyzed (Participants) | 2 | 2 | 2
  48 hour postdosing | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: From 4mL dose administration date to end of the study, approximately 3-5 months for each participant.
Arm/Group | 4 mL | 16 mL | 32 mL
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/13 | 3/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mL (N=13) | 16 mL (N=12) | 32 mL (N=12)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT03408899/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03408899/SAP_001.pdf